CLINICAL TRIAL: NCT01263561
Title: Prospective Randomized Study Comparing Ex-PRESS to Trabeculectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Yvonne Buys, MD, FRCSC; Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0888-A
Record Dates: First submitted 2010-12-14; First posted 2010-12-20 (Estimated); Results first posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Glaucoma
Keywords: glaucoma; filtration surgery; trabeculectomy; ExPRESS shunt
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- trabeculectomy (Active Comparator): trabeculectomy filtering surgery
  Interventions: Procedure: trabeculectomy
- ExPRESS (Experimental): ExPRESS miniature glaucoma drainage device
  Interventions: Procedure: ExPRESS shunt

INTERVENTIONS:
Procedure: ExPRESS shunt — ExPRESS miniature glaucoma drainage device
  Arms: ExPRESS
Procedure: trabeculectomy — trabeculectomy filtering surgery
  Arms: trabeculectomy

SUMMARY:
Prospective randomized study comparing guarded Ex-PRESS to trabeculectomy. Primary outcome: IOP and success (complete success defined as IOP between 5-18 mmHg and 20% reduction from baseline without medication or additional glaucoma surgery and qualified success defined as IOP between 5-18 mmHg and 20% reduction from baseline with or without glaucoma medication but no additional glaucoma surgery). Secondary outcomes: number of glaucoma medications, visual acuity, number of complications, corneal pachymetry and corneal endothelial cell counts.

DETAILED DESCRIPTION:
Complications will be evaluated for the intra-operative, early post-operative (up until 1 month) and late post-operative (from 1 month to 1 year) periods. In addition complications will be evaluated as severe (defined as a permanent reduction in vision or complications requiring a surgical intervention) and not severe (complications which resolve with conservative management). As an individual subject may have more than one complication, the number of complications will be compared between the two surgical groups.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 85
* open-angle glaucoma uncontrolled medically
* intraocular pressure ≥ 18 mmHg
* trabeculectomy as the planned surgical procedure

Exclusion Criteria:

* any previous ocular incisional surgery with the exception of previous clear
* cornea cataract surgery
* uveitis
* vitreous present in anterior chamber
* patient unwilling or unable to accept randomization or to give consent or to attend the follow up visits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham E Trope, Professor, Study Director — University of Toronto; Yvonne M Buys, Professor, Study Director — University of Toronto
Locations (1):
- Department of Ophthalmology and Vision Sciences Toronto Westarn Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740
- [Derived] Gonzalez-Rodriguez JM, Trope GE, Drori-Wagschal L, Jinapriya D, Buys YM. Comparison of trabeculectomy versus Ex-PRESS: 3-year follow-up. Br J Ophthalmol. 2016 Sep;100(9):1269-73. doi: 10.1136/bjophthalmol-2015-307161. Epub 2015 Dec 16. PMID 26674779

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trabeculectomy | ExPRESS
Started | 31 | 33
Completed | 30 | 31
Not Completed | 1 | 2
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trabeculectomy | ExPRESS | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (11.5) | 62 (13.9) | 63.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 21 | 20 | 41
intraocular pressure [Mean (Standard Deviation); unit: mmHg] | 22 (6.8) | 22.6 (10.2) | 22.3 (8.6)
glaucoma medications [Mean (Standard Deviation); unit: number of medications] | 3.4 (1.3) | 3.5 (.9) | 3.5 (1.1)
visual acuity [Mean (Standard Deviation); unit: logMAR] | .48 (.6) | .42 (.6) | .44 (.56)

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Time Frame: 1 year post surgery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Trabeculectomy | ExPRESS
Number analyzed (Participants) | 30 | 31
mmHg | 10.7 (3.5) | 11.2 (4.3)
Statistical Analysis 1: Comparison: Trabeculectomy vs ExPRESS; Test type: Non-Inferiority or Equivalence — A sample size calculation determined that 52 eyes were required to detect a 2.0 mmHg IOP difference with a power of 80%; p = .85, t-test, 2 sided

2. Primary Outcome: Success Rate (IOP Between 5-18 mmHg and 20% Reduction From Baseline) Without Glaucoma Medication
Time Frame: 1 year post surgery
Measure: Number; unit: percentage of participants
Arm/Group | Trabeculectomy | ExPRESS
Number analyzed (Participants) | 30 | 31
percentage of participants | 57 | 71
Statistical Analysis 1: Comparison: Trabeculectomy vs ExPRESS; Test type: Non-Inferiority or Equivalence — Power calculation only for main outcome measure of IOP; p = .24, Kaplan Meier

3. Secondary Outcome: Complications
Description: Complications will be evaluated for the intra-operative, early post-operative (up until 1 month) and late post-operative (from 1 month to 1 year) periods. In addition complications will be evaluated as severe (defined as a permanent reduction in vision or complications requiring a surgical intervention) and not severe (complications which resolve with conservative management). As an individual subject may have more than one complication, the number of complications will be compared between the two surgical groups.
Time Frame: 1 year post surgery
Measure: Number; unit: participants
Arm/Group | Trabeculectomy | ExPRESS
Number analyzed (Participants) | 31 | 33
participants
  Early transient hypotony | 12 | 13
  Late transient hypotony | 2 | 3
  encapsulated bleb | 1 | 0
  choroidal effusion | 1 | 0
  early bleb leak | 2 | 3
  membrane over ExPRESS | 0 | 1
  ExPRESS eroding through sclera | 0 | 1
  Total # of subjects with a complication | 16 | 15
Statistical Analysis 1: Comparison: Trabeculectomy vs ExPRESS; Test type: Non-Inferiority or Equivalence — Power calculation only performed for main outcome measure of IOP; p = 0.80, Chi-squared — Above p is for number of subjects with any complication. P values above 0.05 are considered statistically insignificant in this study

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Trabeculectomy | ExPRESS
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No